CLINICAL TRIAL: NCT06844214
Title: A Phase 1/Phase 2 Open-label Single Arm Study With Dose Escalation (Part A), and Dose Expansion (Part B) Parts to Evaluate the Safety, Tolerability, and Efficacy of SAR446268, an Adeno-associated Viral Vector-mediated Gene Therapy in Participants 10 to 50 Years Old With Non-congenital Myotonic Dystrophy Type 1
Brief Title: A Study to Investigate the Safety, Tolerability, and Efficacy of SAR446268, an Adeno-associated Viral Vector-mediated Gene Therapy in Participants Aged 10 to 50 Years of Age With Non-congenital Myotonic Dystrophy Type 1
Acronym: BrAAVe
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DFI17808; U1111-1290-9594 (Registry Identifier: ICTRP)
Record Dates: First submitted 2025-02-19; First posted 2025-02-25 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Myotonic Dystrophy
MeSH Terms: conditions — Myotonic Dystrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SAR446268 (Experimental): Participants will receive a single dose of SAR446268 on Day 1
  Interventions: Biological: SAR446268

INTERVENTIONS:
Biological: SAR446268 — Pharmaceutical form: Solution for infusion; Route of administration: IV infusion

SUMMARY:
This is a Phase 1/Phase 2 open-label single arm, multicenter, and multinational study with SAR446268 for treatment of male and female participants 10 to 50 years old with non-congenital myotonic dystrophy (DM) type 1 (DM1).

The purpose of this study is to evaluate the safety and efficacy of SAR446268 in knocking down dystrophia myotonica protein kinase (DMPK) messenger ribonucleic acid (mRNA) levels and improving neuromuscular function in DM1 participants receiving a single intravenous (IV) administration of SAR446268. The study consists of a dose escalation part (Part A) during which single ascending doses of SAR446268 will be evaluated in 3 distinct cohorts and an optional 4th dose cohort. Once a safe and effective dose is identified, additional participants will be treated in Part B, the dose expansion phase of the study.

The study duration will be 110 weeks (approximately 2 years) for each participant in Parts A and B respectively and includes a 6-week screening phase and a 104-week follow-up period post-SAR446268 administration.

DETAILED DESCRIPTION:
Each participant meeting the eligibility criteria for each of the study parts will receive a single dose administration of SAR446268.

ELIGIBILITY:
Inclusion Criteria: Participants are eligible to be included in the study only if all of the following criteria apply:

* For Part A, participants must be 18 to 50 years of age inclusive, at the time of signing the informed consent.
* For Part B, participants must be as follows:

  * 10 to 17 years of age inclusive, at the time of signing the informed consent or,
  * 18 to 50 years of age inclusive, at the time of signing the informed consent.
* Participants with non-congenital onset DM1
* Participants presenting with signs of DM1 including myotonia and muscle weakness, as diagnosed previously by a clinician based on medical history.
* Participants with genetic diagnosis of DM1 [cytosine-thymine-guanine (CTG) repeat length ≥50 in one allele from medical history]
* Participants who can walk independently for at least 10 meters at screening (orthoses and ankle braces allowed).
* Participants who have been classified according to cardiac risk by the Investigator as:

  * Moderate risk participants with pacemaker and/or implantable cardioverter-defibrillator (ICD) for Part A
  * Low, moderate, or high cardiac risk for Part B

Exclusion Criteria: Participants are excluded from the study if any of the following criteria apply:

* Participants with neutralizing antibodies against the AAV.SAN011 capsid
* Participants with left ventricular ejection fraction (LVEF) <50%
* Participants with liver or biliary disease defined as having at least one of the following:

  * Alanine aminotransferase (ALT) >2 x ULN and aspartate aminotransferase (AST) >2 x ULN
  * Alkaline phosphatase >2 x ULN
  * Total bilirubin >1.5 x ULN (unless has a genetically confirmed diagnosis of Gilbert's syndrome)
  * Direct bilirubin ≥1.5 x ULN
  * Participants with International normalized ratio >1.5
* Participants with renal disease defined as:

  • Serum creatinine >1.5 x ULN and/or estimated glomerular filtration rate <60 mL/min/1.73 m2 as determined by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) (2021) for those age ≥18 years and Bedside Schwartz Equation for those <18 years
* Participants with chronic respiratory insufficiency and on non-invasive ventilatory support, nighttime ventilatory support or full-time ventilation.
* Participants with contraindication to corticosteroid or with conditions that could worsen in the presence of corticosteroids, as determined by the Investigator.
* Participants with active hepatitis B or C infection; HBsAg (+), or HCV RNA (+), or current antiviral therapy for either.
* Participants with HBcAb (+) who are not amenable for prophylactic anti-HBV therapy or pre-emptive therapy guided by serial HBV DNA monitoring during the corticosteroids therapy.
* Participants at high risk for tuberculosis reactivation during the corticosteroids therapy as determined by the Investigator.
* Participants with a known HIV infection
* Participants with serious intercurrent illness that, in the opinion of the Investigator, would preclude participation in the study or potentially decrease survival.
* Participants with recent history of or current drug or alcohol abuse in the past 12 months prior to screening.
* Participants with history of tibialis anterior biopsy within 12 weeks from Day 1 or planning to undergo tibialis anterior biopsies during the duration of this clinical trial.
* Participants with significant developmental delay, intellectual disability, or behavioral neuropsychiatric manifestations as determined by the Investigator.
* Participants with previous systemic corticosteroids treatment at doses of >5 mg/day within 15 days of Day 1
* Participants with previous treatment with anti-myotonic medication within 15 days of Day 1
* Participants not suitable for participation, whatever the reason, as judged by the Investigator, including medical or clinical conditions, or participants potentially at risk of noncompliance to study procedures.

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 10 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-07-23 (Actual); Primary Completion 2029-02-28 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Part A and Part B: Incidence of treatment-emergent adverse events (TEAEs) following SAR446268 administration | Baseline to Week 52
  Number of TEAEs post-SAR446268 administration
Part B: Proportion of participants with at least 40% DMPK mRNA knockdown in muscle biopsy at Weeks 12 and 52 following SAR446268 administration | Weeks 12 and 52

SECONDARY OUTCOMES:
Part A: Change in 10-meter walk-run test from baseline to Weeks 26 and 52 following SAR446268 administration | Baseline to Week 26 and 52
  The 10-meter walk-run test is a mobility test that measures how fast a participant can traverse 10 meters with or without assisted devices.
Part A: Change in myotonia from baseline to Weeks 26 and 52 following SAR446268 administration as measured by the hand opening time (middle finger) | Baseline to Week 26 and 52
  This test for myotonia measures how quickly a participant can open his/her hand after making a tight fist.
Part A: Change in bilateral hand grip test from baseline to Weeks 26 and 52 following SAR446268 administration | Baseline to Week 26 and 52
  This test for strength of the hand muscles measures the maximum force generated by a participant's hand grip using a dynamometer.
Part A: Proportion of participants with at least 40% DMPK mRNA knockdown in muscle biopsy at Weeks 12 and 52 following SAR446268 administration | Weeks 12 and 52
Part A: Change in DMPK mRNA levels in muscle biopsy from baseline to Weeks 12 and 52 following SAR446268 administration | Baseline to Week 12 and 52
Part A: Change in RNA splicing index in muscle biopsy from baseline to Weeks 12 and 52 following SAR446268 administration | Baseline to Week 12 and 52
Part A: Assessment of the duration of AAV vector shedding of SAR446268 in sampling of urine, saliva, and semen at 4-week intervals following SAR446268 administration | Baseline, Weeks 4, 8, and 12
Part B: Change in 10-meter walk-run test from baseline to Weeks 26 and 52 following SAR446268 administration | Baseline to Week 26 and 52
  The 10-meter walk-run test is a mobility test that measures how fast a participant can traverse 10 meters with or without assisted devices.
Part B: Change in myotonia from baseline to Weeks 26 and 52 following SAR446268 administration as measured by the hand opening time (middle finger) | Baseline to Week 26 and 52
  This test for myotonia measures how quickly a participant can open his/her hand after making a tight fist.
Part B: Change in bilateral hand grip test from baseline to Weeks 26 and 52 following SAR446268 administration | Baseline to Week 26 and 52
  This test for strength of the hand muscles measures the maximum force generated by a participant's hand grip using a dynamometer.
Part B: Change in DMPK mRNA knockdown in muscle biopsy from baseline to Weeks 12 and 52 following SAR446268 administration | Baseline to Week 12 and 52
Part B: Change in RNA splicing index in muscle biopsy from baseline to Weeks 12 and 52 following SAR446268 administration | Baseline to Week 12 and 52
Part B: Assessment of the duration of AAV shedding of SAR446268 in sampling of urine, saliva, and semen at 4-week intervals following SAR446268 administration | Baseline, Weeks 4, 8, and 12

CONTACTS AND LOCATIONS:
Locations (8):
- United States (3):
  - University of Florida, 2004 Mowry Road - Site Number: 8400005, Gainesville, Florida
  - University of South Florida - Neuromuscular Research, 13330 USF Laurel Drive - Site Number: 8400001, Tampa, Florida
  - Columbia University Medical Center - Neurological Institute, 710 W. 168th, 2nd floor, suite 204 - Site Number : 8400003, New York, New York
- Hospital Italiano de Buenos Aires, Juan Domingo Peron 4190 - Site Number: 0320001, Buenos Aires, Argentina
- Investigational Site Number : 0360001, Brisbane, Queensland, Australia
- The Montreal Neurological Institute and Hospital, 3801 rue University - Site Number: 1240001, Montreal, Quebec, Canada
- Investigational Site Number : 3760002, Ramat Gan, Israel
- Investigational Site Number : 8260002, Newcastle upon Tyne, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: DFI17808 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=26793&tenant=MT_SNY_9011